CLINICAL TRIAL: NCT02443402
Title: Sitagliptin for the Prevention and Treatment of Stress Hyperglycemia in Non-Diabetic Patients Undergoing Cardiac Surgery
Brief Title: Sitagliptin in Non-Diabetic Patients Undergoing Cardiac Surgery
Acronym: SITACABG NonDM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00080209
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Results first posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Coronary Artery Disease
Keywords: Non diabetic hyperglycemia
MeSH Terms: conditions — Coronary Artery Disease | interventions — Sitagliptin Phosphate; Insulin; Insulin Glargine; Insulin Lispro; Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitagliptin (Experimental): Subjects undergoing cardiac surgery with no history of diabetes and with normal blood glucose (BG) will be randomized to take sitagliptin. Subjects with stress hyperglycemia (defined as a BG >180 mg/dL) in the intensive care unit (ICU) will continue to receive sitagliptin and will be started on continuous intravenous insulin (Regular Human Insulin) adjusted to achieve and maintain a BG target between 110 - 180 mg/dL following standard hospital protocol. Additionally, once moved to the regular floors and out of ICU, the subjects can receive insulin glargine, insulin lispro, and/or insulin aspart depending on the blood glucose level.
  Interventions: Drug: Sitagliptin; Drug: Regular Human Insulin; Drug: Insulin glargine; Drug: Supplemental insulin (Insulin lispro); Drug: Supplemental insulin (Insulin aspart)
- Placebo (Placebo Comparator): Subjects undergoing cardiac surgery with no history of diabetes and with normal blood glucose (BG) will be randomized to take a placebo. Subjects with stress hyperglycemia (defined as a BG >180 mg/dL) in the intensive care unit (ICU) will continue to receive a placebo and will be started on continuous intravenous insulin (Regular Human Insulin) adjusted to achieve and maintain a BG target between 110 - 180 mg/dL following standard hospital protocol. Additionally, once moved to the regular floors and out of ICU, the subjects can receive insulin glargine, insulin lispro, and/or insulin aspart depending on the blood glucose level.
  Interventions: Drug: Placebo; Drug: Regular Human Insulin; Drug: Insulin glargine; Drug: Supplemental insulin (Insulin lispro); Drug: Supplemental insulin (Insulin aspart)

INTERVENTIONS:
Drug: Sitagliptin — Subjects will take one pill daily until the day prior to them being discharged from the hospital. Sitagliptin will be dispensed orally at 100 mg/day and at a lower dose 50 mg for patients with glomerular filtration rate (GFR) < 30-50. If the calculated GFR drops to 30 mL/min/1.73m2 or below, patients will receive study medication 25mg daily
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Placebo — One pill daily until discharge
  Arms: Placebo
Drug: Regular Human Insulin — Continuous intravenous insulin given to ICU patients with a BG > 180 mg/DL for two consecutive readings and will be started on Regular Human Insulin adjusted to achieve and maintain a BG target between 110 - 180 mg/dL following standard hospital protocol. Intravenous insulin infusion will be continued until the patient is able to eat and/or transferred to non-ICU service. In previous studies, average length of insulin infusion in patients with stress hyperglycemia was 16.9±19 hours and the amount of IV insulin requirement was 18.6±24.3 U/day.
  Other Names: Novolin-R, Humulin-R
Drug: Insulin glargine — When regular insulin is discontinued, if needed, insulin glargine will be given once daily. Patients who required continuous insulin infusion at an average rate >2U/h will be transitioned to basal (to be given approx. 4 hours prior to discontinuing the insulin drip) starting at a dose 0.2 U/Kg/d.
  Subjects with a BG at 140-200 mg/dL will start glargine at 0.2 U/kg weight per day. And subjects with BG between 201-400 mg/dL will start glargine at 0.2 U/Kg/day
  The basal insulin dose will be adjusted as follow:
  * If fasting and pre-dinner BG is between 100 - 180 mg/dL in the absence of hypoglycemia the previous day: no change
  * If fasting and pre-dinner BG is between 180 - 240 mg/dL in the absence of hypoglycemia: increase glargine by 10% every day
  * If fasting and pre-dinner BG is > 241 mg/dL in the absence of hypoglycemia the previous day: increase glargine dose by 20% every day
  * If fasting and pre-dinner BG is < 100 mg/dL in the absence of hypoglycemia: stop glargine
  Other Names: Lantus (glargine)
Drug: Supplemental insulin (Insulin lispro) — Insulin lispro will be administered before meals in addition to scheduled insulin dose following the supplemental insulin scale protocol. At bedtime, half of supplemental sliding scale insulin starting at BG >240 mg/dL will be given.
  For the subjects receiving supplemental insulin lispro with BG levels greater than 180 mg/dL, then supplemental insulin scale is as follows:
  * BG between 181-220 mg/dL; 2-4 units of insulin lispro
  * BG between 221-260 mg/dL; 3-5 units of insulin lispro
  * BG between 261-300 mg/dL; 4-6 units of insulin lispro
  * BG between 301-350 mg/dL; 5-7 units of insulin lispro
  * BG between 351-400 mg/dL; 6-8 units of insulin lispro
  * BG > 400 mg/dL; 7-9 units of insulin lispro
  Other Names: Humalog
Drug: Supplemental insulin (Insulin aspart) — Insulin aspart will be administered before meals in addition to scheduled insulin dose following the supplemental insulin scale protocol. At bedtime, half of supplemental sliding scale insulin starting at BG >240 mg/dL will be given.
  For the subjects receiving supplemental insulin aspart with BG levels greater than 180 mg/dL, then supplemental insulin scale is as follows:
  * BG between 181-220 mg/dL; 2-4 units of insulin aspart
  * BG between 221-260 mg/dL; 3-5 units of insulin aspart
  * BG between 261-300 mg/dL; 4-6 units of insulin aspart
  * BG between 301-350 mg/dL; 5-7 units of insulin aspart
  * BG between 351-400 mg/dL; 6-8 units of insulin aspart
  * BG > 400 mg/dL; 7-9 units of insulin aspart
  Other Names: Novolog

SUMMARY:
The purpose of this study is to compare sitagliptin and placebo for the prevention of high blood glucose during surgery.

DETAILED DESCRIPTION:
About 80% of patients develop high glucose after cardiac surgery. High glucose is linked to an increased risk of hospital complications. High glucose increases the risk of wound infection, kidney failure and death. Patients with high glucose are treated with insulin given through an arm vein or by frequent insulin injections under the skin. This study will determine if sitagliptin can prevent the development of high glucose after heart surgery. Sitagliptin is a diabetes pill approved by the Food and Drug Administration (FDA) to treat patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 18 and 80 years undergoing, cardiac surgery
* No previous history of diabetes
* No previous history of hyperglycemia

Exclusion Criteria:

* Patients with hyperglycemia (blood glucose > 125 mg/dL); or glycated hemoglobin (HbA1c) > 6.5%; or previous treatment with oral antidiabetic agents or insulin
* Severely impaired renal function (serum creatinine ≥3.0 mg/dL or GFR < 30 mL/min) or clinically significant hepatic failure
* Moribund patients and those at imminent risk of death (brain death or cardiac standstill)
* Subjects with gastrointestinal (GI) obstruction or adynamic ileus or those expected to require GI suction
* Patients with clinically relevant pancreatic or gallbladder disease
* Treatment with oral or injectable corticosteroid
* Mental condition rendering the subject unable to understand the scope, and consequences of the study
* Female subjects who are pregnant or breast feeding at time of enrollment into the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital - Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from four academic hospitals including Emory University Hospital, Emory Midtown Hospital, Emory Saint Joseph's, and Grady Memorial Hospital in Atlanta, Georgia between January 2016 and October 2016.
Pre-assignment Details: Of the 68 participants consented for study participation, seven did not begin study participation after randomization. One participant was a screen failure prior to randomization. All participants that began a study intervention were included in the baseline analysis.
Groups:
- Sitagliptin: Subjects undergoing cardiac surgery with no history of diabetes and with normal blood glucose (BG) were randomized to take sitagliptin.
- Placebo: Subjects undergoing cardiac surgery with no history of diabetes and with normal blood glucose (BG) were randomized to take a placebo.
Period: Overall Study
Arm/Group | Sitagliptin | Placebo
Started | 36 | 31
Completed | 32 | 28
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Screen Failure | 1 | 2

BASELINE CHARACTERISTICS:
Population: The participants included in the baseline analysis were randomized to a study arm and received an intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 32 | 28 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (11) | 64 (9) | 64 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 24 | 23 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 20 | 20 | 40
  African American | 9 | 6 | 15
  Other | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 28 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Stress Hyperglycemic Events in the Intensive Care Unit (ICU)
Description: Number of participants who developed stress hyperglycemia (BG >180 mg/dl) during coronary artery bypass grafting (CABG) or after CABG requiring continuous IV insulin infusion (CII) while in the ICU.
Time Frame: Post-Surgery (Up to 4 Days)
Population: Participants that completed all study assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
Participants | 22 | 25

2. Primary Outcome: Number of Subjects With Persistent Hyperglycemia
Description: Number of subjects with persistent hyperglycemia (2 consecutive fasting and/or premeal BG > 180 mg/dL, or with average daily BG >180 mg/dl) who require insulin glargine (rescue therapy) after discontinuation of continuous intravenous insulin (CII)
Time Frame: Post-Surgery (Up to 10 Days)
Population: Participants that completed all study assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
Participants | 7 | 6

3. Secondary Outcome: Need for Continuous Intravenous Insulin (CII) for Treatment of Hyperglycemia
Description: Number of subjects with hyperglycemia (BG >180 mg/dL) who require CII in the ICU.
Time Frame: Post-Surgery (Up to 4 Days)
Population: Participants that completed all study assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
Participants | 7 | 7

4. Secondary Outcome: Mean Daily Intensive Care Unit (ICU) Blood Glucose (BG) Concentration
Description: The blood glucose levels will be assessed throughout the day using a glucose meter. An average will be calculated. The normal BG range for someone with diabetes is 80-130 mg/dL.
Time Frame: Post-Surgery (Up to 4 Days)
Population: Participants that completed all study assessments.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
mg/dL | 137 (16) | 138 (25)

5. Secondary Outcome: Mean Amount of Insulin Therapy in the Intensive Care Unit (ICU)
Description: The mean number of insulin infusions given per day (unit/day) while subjects are in the ICU. The more insulin given, the more hyperglycemic events experienced.
Time Frame: Post-Surgery (Up to 4 Days)
Population: Participants that completed all study assessments.
Measure: Mean (Standard Deviation); unit: units per day
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
units per day | 37 (60) | 83 (64)

6. Secondary Outcome: Duration of Continuous Intravenous Insulin (CII)
Description: Mean number of hours on continuous intravenous insulin (CII) after ICU discharge.
Time Frame: Post-Intensive Care Unit (ICU) Discharge (Up to 4 Days)
Population: Participants that completed all study assessments.
Measure: Mean (Inter-Quartile Range); unit: hours
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
hours | 12 [5 to 88] | 17 [9 to 80]

7. Secondary Outcome: Mean Units Subcutaneous (SQ) Insulin Required
Description: Mean number of supplemental insulin units (lispro or aspart) administered after receiving insulin glargine (SQ insulin).
Time Frame: Post-Surgery (Up to 10 Days)
Population: Participants that completed all study assessments.
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
units | 2.4 (.5) | 2.4 (.9)

8. Secondary Outcome: Mean Blood Glucose (BG) Concentration After Transition From Intensive Care Unit (ICU)
Description: The blood glucose levels will be assessed throughout the day using a glucose meter after transition form the ICU. The normal BG range for someone with diabetes is 80-130 mg/dL.
Time Frame: Post-Surgery (Up to 4 Days)
Population: Participants that completed all study assessments.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
mg/dl | 123 (13) | 124 (16)

9. Secondary Outcome: Total Insulin Therapy in the Intensive Care Unit (ICU)
Description: Total amount of insulin glargine insulin (units) administered in the ICU per day.
Time Frame: Post-Surgery (Up to 4 Days)
Population: Participants that completed all study assessments.
Measure: Mean (Standard Deviation); unit: units per day
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
units per day | 0 (0) | 0 (0)

10. Secondary Outcome: Number of Participants With Severe Hyperglycemic Events During Continuous Insulin Infusion (CII)
Description: Number of participants with two consecutive blood glucose concentrations >180 mg/dL in ICU during CII.
Time Frame: Post-Surgery (Up to 4 Days)
Population: Participants that completed all study assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
Participants | 7 | 6

11. Secondary Outcome: Number of Participants With Hyperglycemia After Transition From Intensive Care Unit (ICU)
Description: Number of participants with blood glucose (BG) >180 after transition from ICU.
Time Frame: Post-Surgery (Up to 10 Days)
Population: Participants that completed all study assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
Participants | 8 | 8

12. Secondary Outcome: Number of Participants With Hypoglycemia During Intensive Care Unit (ICU) Stay
Description: Number of participants with blood glucose (BG) <70 during ICU stay.
Time Frame: Post-Surgery (Up to 4 Days)
Population: Participants that completed all study assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
Participants | 2 | 1

13. Secondary Outcome: Number of Participants With Hypoglycemia After Transition From Intensive Care Unit (ICU)
Description: Number of participants with blood glucose (BG) <70 after transition from ICU.
Time Frame: Post-Surgery (Up to 4 Days)
Population: Participants that completed all study assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
Participants | 1 | 0

14. Secondary Outcome: Number of Participants With Blood Glucose Less Than 40 mg/dl
Description: Number of participants with blood glucose (BG) <40 throughout the duration of hospitalization.
Time Frame: Duration of Hospitalization (Up to 30 Days)
Population: Participants that completed all study assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
Participants | 0 | 0

15. Secondary Outcome: Hospital Mortality Rate
Description: The total number of subject deaths during hospital stay will be recorded.
Time Frame: Post-Surgery (Up to 10 Days)
Population: Participants that completed all study assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
Participants | 0 | 0

16. Secondary Outcome: Intensive Care Unit (ICU) Mortality Rate
Description: The total number of subject deaths during ICU stay will be recorded.
Time Frame: Post-Surgery (Up to 4 Days)
Population: Participants that completed all study assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
Participants | 0 | 0

17. Secondary Outcome: Number of Participants With Cerebrovascular Events
Description: Number of participants that experienced permanent stroke and reversible ischemic neurologic deficit events.
Time Frame: Post-Hospital Discharge (Up to 10 Days)
Population: Participants that completed all study assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
Participants | 2 | 1

18. Secondary Outcome: Hospital Complication Rate
Description: The total number of all complications experienced during hospitalization. Participants may experience more than one complication during hospitalization and these will be included in the hospital complication rate.
Time Frame: Duration of Hospitalization (Up to 30 days)
Population: Participants that completed all study assessments.
Measure: Number; unit: number of complications
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
number of complications | 47 | 57

19. Secondary Outcome: Length of Stay: Intensive Care Unit (ICU)
Description: Number of days in the ICU after coronary artery bypass graft surgery (CABG).
Time Frame: Post-Surgery (Up to 4 Days)
Population: Participants that completed all study assessments.
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
days | 2 [1 to 4] | 2 [1 to 3]

20. Secondary Outcome: Length of Hospital Stay After Study Randomization
Description: Number of days in the hospital after a participant is randomized to a study intervention.
Time Frame: Post-Randomization (Up to 9 days)
Population: Participants that completed all study assessments.
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
days | 6.0 [5.0 to 9.0] | 6.5 [4.5 to 8.0]

21. Secondary Outcome: Number of Participants Re-admitted to the Hospital Due to Wound Infections
Description: Number of subjects readmitted to the hospital within 30 days due to wound infection.
Time Frame: Post-Hospital Discharge (Up to 30 Days)
Population: Participants that completed all study assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
Participants | 1 | 1

22. Secondary Outcome: Number of Participants Re-admitted to the Hospital Not Due to Wound Infections
Description: Number of subjects readmitted to the hospital within 30 days for all causes excluding wound infection.
Time Frame: Post-Hospital Discharge (Up to 30 Days)
Population: Participants that completed all study assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
Participants | 3 | 0

23. Secondary Outcome: Number of Participants With Emergency Room (ER) Visits
Description: Number of subjects returning to the ER up to 30 days (all-cause) after hospital discharge.
Time Frame: Post-Hospital Discharge (Up to 30 Days)
Population: Participants that completed all study assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
Participants | 2 | 1

24. Secondary Outcome: Number of Participants With Infections Not Requiring Hospital Re-admission
Description: Number of subjects with infections not requiring hospital re-admission within 30 days after hospital discharge.
Time Frame: Post-Hospital Discharge (Up to 30 Days)
Population: Participants that completed all study assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
Participants | 0 | 1

25. Secondary Outcome: Number of Subjects Requiring the Use of Inotropes for Greater Than 24 Hours
Description: The number of subjects requiring the use of inotropes for >24 hours post CABG.
Time Frame: Post-Surgery (Up to 2 Days)
Population: Participants that completed all study assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
Participants | 11 | 7

26. Secondary Outcome: Number of Subjects Requiring Re-intubation
Description: The number of subjects requiring re-intubation after CABG.
Time Frame: Post-Surgery (Up to 2 Days)
Population: Participants that completed all study assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
Participants | 1 | 2

27. Secondary Outcome: Number of Subjects Requiring Re-intubation Within 24 Hours
Description: The number of subjects requiring re-intubation with 24 after CABG.
Time Frame: Post-Surgery (Up to 24 Hours)
Population: Participants that completed all study assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
Participants | 2 | 1

28. Secondary Outcome: Number of Subject Requiring Surgical Re-Intervention
Description: The number of subjects that require surgical re-intervention due to mediastinal exploration and post-operative hemorrhage.
Time Frame: Post-Surgery (Up to 10 Days)
Population: Participants that completed all study assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 32 | 28
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected through hospital discharge (up to 30 days).
Arm/Group | Sitagliptin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/28
Serious Adverse Events (participants affected / at risk) | 9/32 | 7/28
Other Adverse Events (participants affected / at risk) | 22/32 | 15/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=32) | Placebo (N=28)
Stroke (Nervous system disorders) | 2 (2) | 1 (1)
Surgical Site Bleeding (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=32) | Placebo (N=28)
Acute Kidney Injury (Renal and urinary disorders) | 5 (5) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 10 (10) | 9 (9)
Ventricular Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Heart Failure (Cardiac disorders) | 2 (2) | 2 (2)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes